CLINICAL TRIAL: NCT00451737
Title: Correlation of 6-Minute Walk Test and Neuromuscular Parameters in the Elderly: Knee Proprioception, Standing Balance, Quadriceps Muscle Strength, Endurance, and Torque Acceleration Energy
Brief Title: Correlation of 6-Minute Walk Test and Neuromuscular Parameters in the Elderly
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9461712111
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2006-01

CONDITIONS: Healthy
Keywords: Six-minute walk test; Neuromuscular system; Influence factors

INTERVENTIONS:
Device: Isokinetic test

SUMMARY:
The six-minute walk test had been used to assessment the cardiopulmonary parameter in patients with lung and heart disease. And it has good reliability and validity. It has been used extensively in research into the aerobic capacity in patients of peripheral vascular disease, neural system disease, and even the muscular-skeletal system disease, such as osteoarthritis, total hip or knee arthroplasty. There were studies investigate the predictors based on cardiopulmonary factors, neuromuscular and skeletal factors of the six-minute walk distance. But the last is the neuromuscular and skeletal factors.

The purpose of this study is to investigate the correlations between the six-minute walk distance and neuromuscular parameters: muscle function (including muscle endurance, muscle strength and muscle power), knee proprioception, and standing balance. For that it could be more useful for evaluation and treatment patients in clinic.

The study was planed to select 100 subjects, they are older than 65 years old with independent walking and without any diagnosis or symptoms about cardiopulmonary or neural disease. The evaluation are including knee proprioception (closed chain, active-active test), six-minute walk test, one leg standing balance test (open and close eyes for 30 seconds), quadriceps muscle strength at velocities of 600/s,1200/s and 1800/s, quadriceps muscle power at 1800/s, and quadriceps muscle endurance.

To investigate the correlations between the six-minute walk distance and characteristics of subjects, the correlations between six-minute walk distance and neuromuscular parameters, including quadriceps muscle function (strength, endurance and power), knee proprioception, and one leg standing balance. And to analyze what's the most contribution to the six-minute walk distance.

ELIGIBILITY:
Inclusion Criteria:

* older than 65 years old
* independent walking

Exclusion Criteria:

* diagnosis or symptoms about cardiopulmonary or neural disease
* depression

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100
Dates: Start 2006-11; Study Completion 2007-03 (Estimated)

PRIMARY OUTCOMES:
six-minute walking test
knee joint reposition test
knee joint muscle strength
ankle joint muscle strength
knee joint muscle endurance
one leg standing balance

CONTACTS AND LOCATIONS:
Overall Officials: Jan Mei Hwa, MS, Study Director — kinesiology laborary of physical therapy in NTU
Locations (1):
- Jan Mei Hwa, Taipei, Taiwan